CLINICAL TRIAL: NCT04125524
Title: Terahertz Metamaterials for Tumour Marker Concentration Identification
Status: Suspended | Type: Observational
Why Stopped: PhD Student completed primary study. Awaiting a new student to take over the project for the secondary objective.
Sponsor: Durham University (Other)
Collaborators: County Durham and Darlington NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 265479
Record Dates: First submitted 2019-10-08; First posted 2019-10-14 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Malignant Tumour
Keywords: Tumour markers
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Surplus serum samples remaining after hospital tests.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Terahertz metamaterials — A diagnostic test used to identify specific tumour markers will be carried out on serum samples using terahertz metamaterials.

SUMMARY:
The research the investigators plan to undertake involves the use of a metamaterial at terahertz frequencies. Serum samples will be tested using the metamaterial to determine if this method can be used to measure the concentration of tumour markers present in the sample. Patients who have been tested for CEA, LDH, CA-125, CA 19-9, CA 15-3, total-hCG and AFP will be used for both the positive and negative samples.

DETAILED DESCRIPTION:
The research the investigators plan to undertake involves the use of a paper substrate with a gold metamaterial on top or a plastic substrate with gold metamaterial on top in physical contact with paper. The metamaterial has an absorption peak within the terahertz frequency range to be investigated (0.75 - 1.1THz). The serum samples will be soaked into the paper fibres which will shift the absorption peak within the terahertz frequency range dependent on the concentration of tumour markers present in the sample. The serum samples will be surplus from samples tested for CEA, LDH, CA-125, CA 19-9, CA 15-3, total-hCG and AFP at the Durham and Darlington NHS Fondation Trust. The samples will be anonymised with the exception of which tumour marker they were tested for and the level measured.

There will be two stages to this research project the initial stage requires 15 samples per proposed marker including 15 samples (across all markers) for negative results. This will be used to identify suitable markers to consider for the second stage. Where 50 to 90 samples of each qualifying marker will be tested dependent on the number required for statistical confidence in stage two with 10 to 18 negative samples required for each qualifying marker, again dependent on the statistical requirements for each marker.

ELIGIBILITY:
Inclusion Criteria:

* Any patient recommended by their health professional to be tested for any of the tumour markers being studied at County Durham and Darlington NHS Foundation Trust for any reason.

Exclusion Criteria:

* Patients with known bloodborne pathogens.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: County Durham and Darlington NHS Foundation Trust
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of detection for any marker | 18 months
  Any correlation showing a difference between samples with marker concentrations above and below the standard threshold values used for tests within the NHS.

SECONDARY OUTCOMES:
Quantifying the quality of detection per marker | 18 months
  Percentage of detectable samples for each specific marker which showed any evidence of detection in outcome 1.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Engineering Durham University, Durham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Outcomes will be shared.